CLINICAL TRIAL: NCT05160987
Title: Effect of Remimazolam With Protocolized Sedation on Critical Ill, Mechanical Ventilated Patients Compared With Midazolam - A Parallel, Multicenter, Single-blind Randomized Controlled Trial
Brief Title: Effect of Remimazolam With Protocolized Sedation on Critical Ill, Mechanical Ventilated Patients Compared With Midazolam
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhujiang Hospital (Other)
Collaborators: Integrated traditional Chinese and Western Medicine Hospital of Southern Medical University (Unknown); First Affiliated Hospital of Shantou University Medical College (Other); Affiliated Hospital of Guangdong Medical University (Other); Yunfu People's Hospital (Unknown); Zhongshan Hospital Of Traditional Chinese Medicine (Other); Guangdong Province Traditional Medical hospital (Unknown); The Third Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Liu Zhanguo, Deputy chief physician of critical medicine department, Zhujiang Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-KY-089-02
Record Dates: First submitted 2021-11-29; First posted 2021-12-16 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Sedation and Analgesia
Keywords: Remimazolam; Midazolam; duration of mechanical ventilation; Sedation
MeSH Terms: conditions — Agnosia | interventions — remimazolam; Midazolam

STUDY DESIGN:
Intervention Model Description: The participants in remimazolam group receive intravenous remimazolam. The participants in midazolam group receive midazolam.
Who Masked: Participant
Masking Description: single-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remimazolam Group (Experimental): The patients are administered with sedation of remimazolam and analgesia of remifentanil on the basis of routine treatment. If the patient does not receive sedative drug before enrollment, patient would be administered with a bolus of remimazolam with 0.1-0.3mg/kg intravenously in 1 minute for the first time. And maintenance dose is 0.25-0.1mg/kg/h, meanwhile the dose of remimazolam should be titrated according to RASS scores. Nonbenzodiazepines could be administrated to the patients if sedation targets were not achieved, and the medication and dosage is recorded.
  Interventions: Drug: Remimazolam
- Midazolam Group (Placebo Comparator): The patients are administered with sedation of midazolam analgesia of remifentanil on the basis of routine treatment. If the patient does not receive sedative drugs before enrollment, patients would be administered with a bolus of midazolam with 0.01-0.05mg/kg intravenously in 1 minute for the first time. And the maintenance dose is 0.02-0.1mg/kg/h, meanwhile the dose of midazolam should be titrated according to RASS scores. Nonbenzodiazepines could be administrated to the patients if sedation targets were not achieved, and the medication and dosage is recorded.
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Remimazolam — Remimazolam will be diluted with 0.9% saline to ensure that the therapeutic drug and placebo are identical in appearance, and 50 ml syringes will serve as the containers for all intravenous drugs.
  Arms: Remimazolam Group
Drug: Midazolam — Midazolam will be diluted with 0.9% saline to ensure that the therapeutic drug and placebo are identical in appearance, and 50 ml syringes will serve as the containers for all intravenous drugs.
  Arms: Midazolam Group

SUMMARY:
In this parallel, multicenter, single-blind randomized controlled trial, mechanical ventilated patients will be randomly assigned to two groups. One receives remimazolam to achieve sedation goals, while the other receives Midazolam. The primary outcome is the effect of remimazolam on duration of mechanical ventilated of critical patients compared to midazolam.

DETAILED DESCRIPTION:
Investigational drug#remimazolam for injection Study title#Effect of Remimazolam with Protocolized Sedation on Critical Ill, Mechanical Ventilated Patients Compared with Midazolam - A parallel, Multicenter, Single-blind Randomized Controlled Trial Principal Investigator#Professor Zhanguo Liu, Dr.Jing Cai, Department of Critical Care Unit, Zhujiang Hospital, Southern Medical University Study subjects#Critical ill patients that are mechanically ventilated within the first 48h of admission to the ICU and who would remain in the ICU for over 72h are enrolled in this study. The ages of patients should be in the range from 18 to 80.

Study phase# Investigator Initiated Trial(IIT) Study objectives#The objective of the study is to determine whether remimazolam, compared with midazolam, reduces duration of ventilation in severe patients.

Study design#A parallel, Multicenter, Single-blind Randomized Controlled Trial. Medication method#Remimazolam group#Patients are administered with a bolus of remimazolam with 0.1-0.3mg/kg intravenously in 1 minute for the first time. And the maintenance dose is 0.25-0.1mg/kg/h, meanwhile the dose of remimazolam should be titrated according to Richmond Agitation Sedation Scale (RASS) scores. Nonbenzodiazepines could be administrated to the patients if sedation targets were not achieved.

Midazolam group#Patients are administered with a bolus of midazolam with 0.01-0.05mg/kg intravenously in 1 minute for the first time. And maintenance dose is 0.02-0.1mg/kg/h, meanwhile the dose of midazolam should be titrated according to Richmond Agitation Sedation Scale (RASS) scores. Nonbenzodiazepines could be administrated to the patients if sedation targets were not achieved.

Spontaneous breathing test (SBT) is conducted daily while patients are stable. Weaning would be considered after a successful SBT, and the sedation for study need to be stopped subsequently. If the weaning failed, mechanical ventilation and sedation would be used immediately according to sedation targets. Weaning success is defined as the ability to successfully complete the SBT and sustain spontaneous breathing for 48h after extubation.

Course#28days Sample size#440. Sites#15 Primary endpoint#Duration of mechanical ventilation(weaning success is typically regarded as consecutive ventilator-free over 24h following liberation from a ventilator. The duration of mechanical ventilation is from the enrollment time to the weaning time. The study and observation would be stopped due to difficult ventilator weaning, which features weaning failure repeatedly for 3 weeks.) Secondary endpoints#

1. Duration of endotracheal intubation(calculated from the time of enrollment);
2. Completion rate of sedation goals (completion rate of sedation goal = days of achieving sedation goals / total days of sedation (days from enrollment to successful ventilator withdrawal) × 100%）)；
3. Sedation remediation is defined as requiring combination with other nonbenzodiazepines sedations.
4. Length of stay in ICU and total length of stay (time from admission to discharge);
5. Others: anterograde amnesia, 28 day mortality, total cost of sedative drugs in ICU, hospitalization expenses in ICU; Anterograde amnesia used a questionnaire that is record to assess the patient's forgetfulness.

Safety endpoints#

1. Incidence of Hypotension(20% fall in systolic pressure).
2. Incidence of Delirium.
3. Incidence of spontaneous extubation.
4. Incidence of reintubation in 12h or tracheotomy.
5. Incidence of Myasthenia.(following weaning from ventilations)
6. Incidence of thrombus.(lower extremity deep venous thrombosis)

ELIGIBILITY:
Inclusion Criteria:

1. Critical ill patients that are mechanically ventilated within the first 48h of admission to the ICU and who would remain in the ICU for over 72h were enrolled in this study.
2. Age 18-80 years.
3. Voluntary informed consent.

Exclusion Criteria:

1. Surgical treatment is performed within 24 hours.
2. Craniocerebral injury, post neurosurgery, non drug coma, mental illness or peripheral neuropathy.
3. Heart rates are less than 50 beats / min or severe atrioventricular block without pacemaker support.
4. The mean arterial pressure is less than 55 mmHg even though fluids and vasoactive drugs are administrated.
5. Patients who are known or suspected allergy to benzodiazepines, propofol, dexmedetomidine or opioids.
6. History of alcohol and drug abuse.
7. End stages of lung diseases, such as pulmonary fibrosis, lung damage, etc.
8. Pregnancy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2022-03-29 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Duration of mechanical ventilation | From the date of enrollment until the date of successful ventilator withdrawal, assessed up to 28 days
  Weaning success is typically regarded as consecutive ventilator-free over 24h following liberation from a ventilator. The duration of mechanical ventilation is from the enrollment time to the weaning time.
  The study and observation would be stopped due to difficult ventilator weaning, which features weaning failure repeatedly for 3 weeks.

SECONDARY OUTCOMES:
Duration of endotracheal intubation | From the date of enrollment until the date of pulling out the endotracheal tube, assessed up to 28 days
  Duration of endotracheal intubation
Completion rate of sedation goal | From the date of enrollment until the date of successful ventilator withdrawal, assessed up to 28 days
  completion rate of sedation goal = days of achieving sedation goals / total days of sedation (days from enrollment to successful ventilator withdrawal) × 100%
Remediation is defined as requiring combination with other sedations | From the date of enrollment until the date of successful ventilator withdrawal, assessed up to 28 days
  If the sedation goal cannot be reached, the clinician will use non benzodiazepines according to the actual situation of the patient, and record the medication and dosage.
Length of stay in ICU and total length of stay | From the date of admission in ICU until the date of transfer from ICU
  Length of stay in ICU and total length of stay
Anterograde amnesia | From the date of enrollment until the date of successful ventilator withdrawal
  Anterograde amnesia used a questionnaire to record their memories of related events during mechanical ventilation (turning over, sputum suction, vascular catheterization, nocturnal nursing medication and other invasive operations). Assess the patient's forgetfulness.
28 day mortality | From the date of enrollment until the date of death from any cause, assessed up to 28 days
  28 day mortality

CONTACTS AND LOCATIONS:
Overall Officials: Zhanguo Liu, M.D.PhD, Principal Investigator — Department of Critical Care Medicine of Zhujiang Hospital
Locations (1):
- Department of Critical Care Medicine of Zhujiang Hospital,Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
Since some data may involve patients privacy. We have no plans to share data so far, and some data may be shared later depending on the patient's wishes.